CLINICAL TRIAL: NCT03802539
Title: 5-year Clinical Evaluation of Cavity Lining on the Restoration of Root Surface Caries Lesions: A Controlled Randomized Clinical Trial
Brief Title: 5-year Clinical Evaluation of Cavity Lining on the Restoration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Uzay Koc, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HEK 11/54-8
Record Dates: First submitted 2019-01-06; First posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Teeth; Lesion; Dental Root Caries
Keywords: Root caries; Cavity lining; Composite resin restorations; Self-etch adhesive
MeSH Terms: conditions — Root Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glass Liner (Experimental): Tooth restoration with a glass ionomer liner material under a nanohybrid composite resin
  Interventions: Device: Glass Liner
- No liner (No Intervention): Tooth restoration without a glass ionomer liner material under a nanohybrid composite resin

INTERVENTIONS:
Device: Glass Liner — restoration of root caries according to two different protocols
  Arms: Glass Liner

SUMMARY:
The purpose of this double-blind, randomized trial is to compare the clinical performance of a composite restorations in root surface carious lesions with or without resin modified glass ionomer lining.

DETAILED DESCRIPTION:
Thirty-nine patients with at least one pair of equivalent root caries lesions and a mean age of 39.6 years (range 18-65 years; median 39 years) were enrolled in this study. After caries removal, the depth, length, and width of the cavity were measured. Lesions in the same patient was randomly divided into two groups, and the dentin surfaces were either lined with resin-modified glass ionomer liner (Glass liner II, Willmann & Pein GmbH Dental, Barmstedt, Germany) or not. All cavities were restored with nanohybrid composite resin (Clearfil Majesty Esthetic, Kuraray, Tokyo, Japan). A total of 100 restorations (50 lined, 50 unlined) were placed according to manufacturer's instructions. The restorations will be evaluated at baseline and at 6, 12, 24, 36, 48 months and 5-year after placement using the modified Haveman Criteria for marginal adaptation, anatomic form, marginal staining, anatomic form, caries in adjacent tooth structure, caries at the cavosurface margin and sensitivity. Statistical analysis will be conducted using the Chi- Square, Fisher's Exact, Mann Whitney-U and Cochran Q tests at a significance level of 5% (P < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Non-hospitalized, healthy patients that were seeking dental treatment for caries lesions on the root surface

Exclusion Criteria:

* Patients who were under the age of 18 years
* Complex medical history
* Severe or chronic periodontitis
* Extreme carious activity
* Heavy bruxism
* Very deep or superficial carious lesions
* Previously restored and abutment teeth

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Retention Outcome | 5 years
  1.Retention Alpha for at least 90% of the restorations The primary factor for determining the clinical performance of a restorative material is the retention rate. It represents the survival rates of the restorations after a period of time. According to ADA (American Dental Association) guidelines, a restorative material should show at leat 90% alpha retention rate after 18 months to be considered as clinically acceptable. The retention is assessed as alpha (retentive restoration) or charlie (failed restoration). Clinical evaluation is performed to examine if the restoration is in place or has fallen.

REFERENCES:
- [Derived] Koc Vural U, Gokalp S, Kiremitci A. Effect of cavity lining on the restoration of root surface carious lesions: a split-mouth, 5-year randomized controlled clinical trial. Clin Oral Investig. 2020 Feb;24(2):979-989. doi: 10.1007/s00784-019-03001-z. Epub 2019 Jul 4. PMID 31273529